CLINICAL TRIAL: NCT06519643
Title: Building Your Successful Nursing Career: Evaluating the Effectiveness of a Career Planning Mobile Application for Male Nurses - a Randomized Double-blind Controlled Trial
Brief Title: Building Your Successful Nursing Career
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Principal Investigator, Hsing-Yi Yu, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D000009238-1
Record Dates: First submitted 2024-07-14; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Nurse's Role; Gender; Professional Burnout
Keywords: male nurse; career plan; mobile application (App); intervention study; randomized controlled trial
MeSH Terms: conditions — Coitus; Burnout, Professional; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The investigators will compare the pre- and post-test differences between the experimental group and the control group. Both the experimental and control groups will fill in the structured questionnaires online at the time before the intervention (Baseline data) and at 0, 6, 12, 18, and 24 months after the intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the effectiveness of a career planning mobile application for male nurses (Experimental): This study aims to evaluate a career planning mobile app specifically tailored for male nurses. The investigators will compare the pre- and post-test differences between the experimental group and the control group. The experimental group will receive the full career planning mobile application intervention, while the control group will receive a sham treatment.
  Interventions: Behavioral: career planning application
- control (Sham Comparator): This study aims to evaluate a career planning mobile app specifically tailored for male nurses. The investigators will compare the pre- and post-test differences between the experimental group and the control group. The experimental group will receive the full career planning mobile application intervention, while the control group will receive a sham treatment.
  Interventions: Behavioral: career planning application

INTERVENTIONS:
Behavioral: career planning application — Arm 1 [Experimental group]: The experimental group will be assigned to participate in a career planning application named "Building Your Successful Nursing Career" App for six months. They will receive the full career planning mobile application intervention along with two online career mentoring sessions.
  Arm 2 [Control group]: The control group will also be assigned to participate in a career planning application named "Building Your Successful Nursing Career" App for six months. However, the control group will only receive a sham treatment. They will only access a few interfaces of the app.

SUMMARY:
This study aims to evaluate a career planning mobile App specifically tailored for male nurses.This three-year experimental project aims to recruit 120 male nurses (60）in the experimental group and 60 in the control group). Employing a prospective double-blind randomized controlled trial (RCT) design, the study will include six follow-up points (pre-intervention, post-intervention at 0, 6, 12, 18, and 24 months) to examine the effectiveness of career self-efficacy, career adaptive behaviors, occupational resilience, career success, and career continuity intentions of male nurses over time. The repeated measures data will be analyzed with the intention-to-treat analysis method and General Estimating Equations (GEE). This research represents an innovative development of the world's first theoretically grounded career planning mobile App for male nurses.The study's results can serve as a valuable reference for future career planning initiatives in nursing practice and education.

DETAILED DESCRIPTION:
This study is a longitudinal study that adopts a double-blind randomized controlled trial (RCT). The study will recruit 120 male nurses and allocate them into the intervention group and the control group in a 1:1 ratio (60 in each group). Based on Super's (1957) career development theory and the four-stage career classification, the participating male nurses will be divided into the exploration stage (experience ≤ 2 years), establishment stage (experience 2-5 years), and maintenance stage (experience 5-15 years), with career stage as a confounding factor. The study uses 1:1:1 stratified randomization to ensure that the number of cases in the experimental group (n=60, exploration stage: establishment stage: maintenance stage = 20:20:20) and the control group (n=60) is the same, as well as the homogeneity of the career stage variables of the two groups. All included subjects will undergo an online pre-test (T0) before allocation, and then enter the experimental group or the control group according to the random assignment results. Both groups will be invited to use the "Building Your Successful Nursing Career" App for six months, with the experimental group receiving the full career planning mobile application intervention and two online Career Mentoring Programs, while the control group receives a sham treatment. Both groups will undergo five follow-up online data collections (0, 6, 12, 18, and 24 month post-intervention). The effectiveness of the career planning mobile application intervention on male nurses' career self-efficacy, career adaptive behaviors, occupational resilience, career success, and career continuity intentions will be examined using the intention-to-treat analysis method and General Estimating Equations (GEE).

ELIGIBILITY:
Inclusion Criteria:

1. Male nursing staff currently engaged in clinical nursing work.
2. Care Within 15 years of working experience.
3. Have a mobile phone with Internet access.
4. Have clear consciousness and can understand and answer the researcher's questions.
5. Audible and understandable Or understand Chinese.
6. Willing to participate in this study and sign the subject consent form.

Exclusion Criteria:

1. Unwilling to participate in this study.
2. Those who cannot download the App.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-05 (Estimated)

PRIMARY OUTCOMES:
career self-efficacy | before intervention and 0, 6, 12, 18, and 24 months post-intervention
  career self-efficacy will be collected by online structure questionnaire
career adaptive behaviors | before intervention and 0, 6, 12, 18, and 24 months post-intervention
  career adaptive behavior will be collected by online structure questionnaire
occupational resilience | before intervention and 0, 6, 12, 18, and 24 months post-intervention
  occupational resilience will be collected by online structure questionnaire
career success | before intervention and 0, 6, 12, 18, and 24 months post-intervention
  career success will be collected by online structure questionnaire
career continuity intentions | before intervention and 0, 6, 12, 18, and 24 months post-intervention
  career continuity intentions will be collected by online structure questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chao Yi-Ping, PhD, Study Director — Chang Gung University; Chiang Yueh-Tao, PhD, Study Director — Chang Gung University; DAI HUNG -DA, PhD, Study Director — Taipei Veterans General Hospital, Taiwan; Shen Yung-Chao, M.S., Study Director — New Taipei Municipal Tu-Cheng Hospital; Lou Jiunn-Horng, PhD, Study Director — Hsin Sheng College of Medical Care and Management

IPD SHARING:
Plan to Share IPD: No